CLINICAL TRIAL: NCT02528279
Title: Prospective Assessment of Relapse Characteristics of Plasmodium Ovale and Antimalarial Treatment Efficacy of Artemether-lumefantrine for Mixed Species and Non-falciparum Malaria in Gabon
Brief Title: Relapses in Plasmodium Ovale and Efficacy of Artemether-lumefantrine for Mixed Species and Non-falciparum Malaria
Acronym: REPLAMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Ramharter, Assoc. Prof., MD, MSc, Albert Schweitzer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Rep001
Record Dates: First submitted 2015-04-28; First posted 2015-08-19 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Plasmodium ovale; relapse; artemether-lumefantrine; mixed species malaria; non-falciparum malaria
MeSH Terms: conditions — Malaria; Recurrence | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coartem (Other): Patients will receive the study drug combination artemether-lumefantrine (Coartem®) orally as a 6 dose regimen for three consecutive days. Tablets are available as a fixed dose combination of 20mg artemether plus 120mg lumefantrine. The dosing will be based on the body weight and follow the manufacturer's recommendations:
  Body weight 5-14kg: 1 tablet; Body weight 15-24kg: 2 tablets; Body weight 25-34kg: 3 tablets; Body weight > 34kg: 4 tablets; The respective amount of tablets is to be taken at hours 0, 8, 24, 36, 48 and 60 with fatty food.
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: Coartem — Patients will receive the study drug combination artemether-lumefantrine (Coartem®) orally as a 6 dose regimen for three consecutive days. Tablets are available as a fixed dose combination of 20mg artemether plus 120mg lumefantrine. The dosing will be based on the body weight and follow the manufacturer's recommendations:
  Body weight 5-14kg: 1 tablet; Body weight 15-24kg: 2 tablets; Body weight 25-34kg: 3 tablets; Body weight > 34kg: 4 tablets; The respective amount of tablets is to be taken at hours 0, 8, 24, 36, 48 and 60 with fatty food.

SUMMARY:
Malaria is a protozoan infection transmitted by anopheline mosquitoes. The most severe forms are caused by Plasmodium (P) falciparum and to a much lesser extent by P. vivax.

Although the interest in research on malaria has increased during the last years, yet little research is conducted on the "neglected" malaria species P. ovale and P. malariae. P. ovale being first described in 1922, it still remains unclear whether it displays dormant pre-erythrocytic liver stages, so called hypnozoites, or not. Primaquine, the only marketed drug with liver stage activity at present, can cause severe hemolysis in glucose-6-phosphate dehydrogenase (G6PD) deficient persons and methemoglobinemia. Because G6PD is widely spread in Central Africa, it is important to explore whether additional intake of liver-active medication is really needed and on this account further research to investigating new treatment options with liver stage activity should be conducted.

While, due to widespread resistance, treatment recommendations for P. falciparum and mixed infections have switched from chloroquine to the safer applicable artemisinin-based combination therapies (ACTs), World Health Organization (WHO) guidelines still suggest chloroquine as first line treatment for P. malariae and P. ovale mono infections. Further studies assessing alternative treatment options are largely missing.

Summing up the current situation for both topics shows the need for further research. Therefore this study aims to assess the evidence and characterize the frequency of relapses in P. ovale infections with respect to differences between its subspecies as well as the effectiveness of the ACT artemether-lumefantrine in P. malariae and P. ovale mono- and mixed infections.

DETAILED DESCRIPTION:
Although P. ovale hypnozoites have never been demonstrated by biological experiments and findings in the literature about relapses are controversial, a 14 days primaquine standard therapy is recommended for every patient suffering from P. ovale infection. As there is no clear evidence of relapses of P. ovale it is of importance to conclusively analyze clinical evidence for its relapse potential to evaluate the necessity for further anti-relapse treatment options.

Moreover, summarizing the actual situation shows the need for further evaluation of the clinical use of ACTs in non-falciparum infections:

* Firstly, molecular diagnostic methods indicate that P. malariae and P. ovale are more prevalent than previously thought. In many settings malaria is treated on clinical suspicion. Diagnosis by microscopy is difficult if parasitemia is low and differentiation of species requires experience. This leads to the assumption that P. malariae and P. ovale infections are already blindly treated with the common ACTs recommended for P. falciparum malaria. The evaluation of artemisinin based combination therapies for non-falciparum malaria is therefore essential.
* Secondly, combination therapies have proven to be protective for the emergence of resistant parasites and in Asia combination therapy could even reduce resistance. As chloroquine-resistant P. malariae parasites have been reported, a combination therapy should be implemented in order to stop the emergence and spread of further resistance. Additionally, artemisinins can, in contrast to chloroquine, reduce transmissibility by their gametocytocidal activity.

A uniform treatment algorithm for all four Plasmodium species would simplify and facilitate treatment of malaria. With the reduction of chloroquine use in settings of poor quality diagnosis, the risk of fatal treatment failure due to wrongly administered chloroquine to chloroquine-resistant P. falciparum would be decreased. Finally, if no 8-aminoquinoline treatment was necessary for P. ovale infections, this could improve the safety and compliance of treatment.

The study is designed as an open label prospective study with a within group design. Patients enrolled will receive oral artemether-lumefantrine tablets as a 6 dose regimen over 3 consecutive days (Day 0, 1 and 2). Dosage depends on the patient's weight is according to the manufacturers recommendations. Patients will be followed for 42 days. If P. ovale is diagnosed at baseline, a one-year follow-up will be conducted every second week.

Parasite density, expressed as the number of parasites per microliter (µl) of blood, will be measured regularly to determine parasite clearance time (PCT).

Blood smears preparation, staining, examination and interpretation will be done according to the Lambaréné method. Thick and thin blood films for parasite count and species diagnosis should be obtained and examined at screening on D0 to confirm inclusion/exclusion criteria. Thick blood films will be examined every 24h following first dose administration and until the parasites have cleared. Thick and thin blood films will be also examined on Days 7, 14, 21, 28, 35 and 42 or on any other day if the patient spontaneously returns. For participants with P. ovale infection at baseline, reading of thick and thin blood films will be continued every second week for up to one year. In case of reappearance of parasites, Coartem will be administered again and Follow-up will be continued as scheduled.

Diagnosis of P. ovale will be effected by PCR. Furthermore, genotyping studies will be used to differentiate a new infection from relapse or recrudescence and to confirm microscopic diagnosis of species. Plasma samples will be collected and stored for further pharmacokinetic analysis 7 days after treatment initiation.

To determine the efficacy clinically, body temperature and clinical signs and symptoms of malaria will be assessed. Safety assessments include physical examination, vital signs and hematology.

Adverse Events and Serious Adverse Events will be ascertained. The investigator or his / her staff will notify the Independent Ethics Committee of all Serious Adverse Events as soon as possible and in accordance with local regulations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 1 year
* Presence of uncomplicated malaria infection confirmed by: fever or history of fever in the previous 3 days, and positive microscopy of P. malariae, P. ovale or mixed infection with parasite density > 10 - 200000/µl of blood
* Residence in vicinity and no travel plans for the next 6 months
* Written informed consent by the patient or the legal representative and where possible, patient assent will be sought. If the patient/parent/guardian is unable to write, witnessed consent is permitted according to local ethical considerations.

Exclusion Criteria:

* Presence of P. falciparum monoinfection
* Presence of severe malaria (clinical WHO criteria)
* Presence of other febrile conditions
* Known history of hypersensitivity, allergic or adverse reactions to artemether or lumefantrine
* Intake of any antimalarials or antibiotics with known antimalarial activity in the past 72 hours
* Intake of an 8-aminoquinoline antimalarial or atovaquone-proguanil in preceding 28 days
* Pregnant women in first trimenon

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response (WHO criteria for antimalarial drug trials) | 28 days
  Adequate clinical and parasitological response on Day 28

SECONDARY OUTCOMES:
Parasite clearance time | 7 days
Fever clearance time | 7 days
Reappearance of P. ovale parasitemia | from day 29 - 2 years of follow up
  Evidence and characterization of duration and frequency of relapses due to Plasmodium ovale after day 28. This is a disctinct outcome measure from the primary outcome and will be presented seperately.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ramharter, Prof., Principal Investigator — Centre de Recherches Médicales de Lambaréné
Locations (2):
- Gabon (2):
  - Centre de Recherches Médicales de Lambaréné, Hôpital Albert Schweitzer, Lambaréné, Moyen-Ogooué Province
  - Centre de Recherches Médicales de Ngounié, Fougamou, Ngouni Province

REFERENCES:
- [Background] Planche T, Krishna S, Kombila M, Engel K, Faucher JF, Ngou-Milama E, Kremsner PG. Comparison of methods for the rapid laboratory assessment of children with malaria. Am J Trop Med Hyg. 2001 Nov;65(5):599-602. doi: 10.4269/ajtmh.2001.65.599. PMID 11716121
- [Background] Richter J, Franken G, Mehlhorn H, Labisch A, Haussinger D. What is the evidence for the existence of Plasmodium ovale hypnozoites? Parasitol Res. 2010 Nov;107(6):1285-90. doi: 10.1007/s00436-010-2071-z. Epub 2010 Oct 5. PMID 20922429
- [Background] Maguire JD, Sumawinata IW, Masbar S, Laksana B, Prodjodipuro P, Susanti I, Sismadi P, Mahmud N, Bangs MJ, Baird JK. Chloroquine-resistant Plasmodium malariae in south Sumatra, Indonesia. Lancet. 2002 Jul 6;360(9326):58-60. doi: 10.1016/S0140-6736(02)09336-4. PMID 12114045
- [Background] Greenwood BM, Bradley AK, Greenwood AM, Byass P, Jammeh K, Marsh K, Tulloch S, Oldfield FS, Hayes R. Mortality and morbidity from malaria among children in a rural area of The Gambia, West Africa. Trans R Soc Trop Med Hyg. 1987;81(3):478-86. doi: 10.1016/0035-9203(87)90170-2. PMID 3318021
- [Background] Perandin F, Manca N, Calderaro A, Piccolo G, Galati L, Ricci L, Medici MC, Arcangeletti MC, Snounou G, Dettori G, Chezzi C. Development of a real-time PCR assay for detection of Plasmodium falciparum, Plasmodium vivax, and Plasmodium ovale for routine clinical diagnosis. J Clin Microbiol. 2004 Mar;42(3):1214-9. doi: 10.1128/JCM.42.3.1214-1219.2004. PMID 15004078
- [Derived] Groger M, Veletzky L, Lalremruata A, Cattaneo C, Mischlinger J, Zoleko-Manego R, Endamne L, Klicpera A, Kim J, Nguyen T, Flohr L, Remppis J, Matsiegui PB, Adegnika AA, Agnandji ST, Kremsner PG, Mordmuller B, Mombo-Ngoma G, Ramharter M. Prospective Clinical Trial Assessing Species-Specific Efficacy of Artemether-Lumefantrine for the Treatment of Plasmodium malariae, Plasmodium ovale, and Mixed Plasmodium Malaria in Gabon. Antimicrob Agents Chemother. 2018 Feb 23;62(3):e01758-17. doi: 10.1128/AAC.01758-17. Print 2018 Mar. PMID 29311086